CLINICAL TRIAL: NCT00244491
Title: The Care Transitions Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The John A. Hartford Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 00-1036
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Continuity of Patient Care
Keywords: care transitions; geriatric; care coordination; self-management; chronic illness; patient-centered care
MeSH Terms: conditions — Chronic Disease

INTERVENTIONS:
Behavioral: Care Transitions Intervention

SUMMARY:
This intervention tests whether encouraging older patients and their caregivers to assert a more active role in their care transitions could improve clinical outcomes. Patients are supported by a nurse transition coach and specific tools, including a Personal Health Record.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this study, patients from the participating delivery system had to: 1) be age 65 years or older, 2) be admitted to one of the participating delivery system's contract hospitals during the study period for a non-psychiatrically-related condition, 3) be community-dwelling (i.e., not from a long-term care facility), 4) reside within a predefined geographic radius of the hospital (thereby making a home visit feasible), 5) have a working telephone, 6) be English-speaking, 7) show no documentation of dementia in the medical record, 8) have no plans to enter hospice, 9) not be participating in another research protocol, and 10) have documented in their medical record at least one of 11 diagnoses, including stroke, congestive heart failure, coronary artery disease, cardiac arrhythmias, chronic obstructive pulmonary disease, diabetes, spinal stenosis, hip fracture, peripheral vascular disease, deep venous thrombosis, or pulmonary embolism.

Exclusion Criteria:

* Those who did not meet the inclusion criteria.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1400
Dates: Start 2002-09; Study Completion 2003-08

PRIMARY OUTCOMES:
Rehospitalization rate at 30, 90 and 180 days after index hospitalization.

SECONDARY OUTCOMES:
Rehospitalization rate at 30, 90 and 180 days after index hospitalization. Rehospitalization for the same condition as the index hospital stay, at 30, 90 and 180 days.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A. Coleman, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States

REFERENCES:
- [Result] Coleman EA, Parry C, Chalmers S, Min SJ. The care transitions intervention: results of a randomized controlled trial. Arch Intern Med. 2006 Sep 25;166(17):1822-8. doi: 10.1001/archinte.166.17.1822. PMID 17000937